CLINICAL TRIAL: NCT00549705
Title: Registry of Hospitalized Patients Treated With Fondaparinux
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Samuel Z. Goldhaber, MD, Brigham and Women's Hospital
Other Study IDs: 2007-P-001294
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Anticoagulation; Thrombosis; Bleeding; Clotting; Pulmonary Embolism; Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Thrombosis; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Registry of Hospitalized patients at Brigham and Women's Hospital treated with Fondaparinux

DETAILED DESCRIPTION:
The use of antithrombotic agents in the hospital is the mainstay of therapy for the treatment or prophylaxis of venous thromboembolism (VTE) and acute coronary syndrome (ACS). Concern with the administration of heparins and risk for adverse sequelae has led to the development of newer, longer-acting agents. Fondaparinux offers once daily administration with only an extremely small risk of developing heparin induced thrombocytopenia.

Recent data have further demonstrated the efficacy and safety of Fondaparinux in VTE and ACS, expanding its use in clinical practice. We aim to: 1) determine how Fondaparinux is being used in a "real life" clinical setting, a tertiary-care academic medical center (BWH), and 2) assess the associated clinical outcomes at 90 days after initiation of Fondaparinux.

ELIGIBILITY:
Inclusion Criteria:

* BWH hospitalized patients receiving Fondaparinux

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: BWH hospitalized patients receiving Fondaparinux
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Venous Thromboembolism and Bleeding Events | 90 Days

SECONDARY OUTCOMES:
Mortality | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- See also: North American Thrombosis Forum (NATF) — http://www.NATFonline.org